CLINICAL TRIAL: NCT02395276
Title: Efficacy of Hypothermia Therapy in Pediatric Cardiac Intensive Care Unit in Children Suspected for Brain Injury
Brief Title: Hypothermia Therapy in Pediatric Cardiac Intensive Care Unit for Suspected for Brain Injury
Acronym: Coolheart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Omer Bar-Yosef, Senior Physician, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMC-0616-13
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Congenital Heart Defects; Brain Ischemia; Hypoxia Brain; Child; Hypothermia, Induced
Keywords: Congenital Heart Defects; Hypoxic Ischemic Brain Injury; Hypothermia Therapy; Pediatrics
MeSH Terms: conditions — Heart Defects, Congenital; Brain Ischemia; Hypoxia, Brain; Hypothermia; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Whole body hypothermia (Active Comparator): Children that had an event suspected for hypoxic ischemic brain injury, according to the inclusion criteria, will be randomly allocated for whole body hypothermia therapy. Treatment will be initiated within 6 hours of the event, the child will be dressed with a cooling suit and their temperature will be monitored. Whole body hypothermia will be to 33 +/- 1 °C . Treatment period will be 48 hours with 24 hours warming up period.
  Interventions: Device: Whole body hypothermia
- Whole body normothermia (Placebo Comparator): Children that had an event suspected for hypoxic ischemic brain injury, according to the inclusion criteria, will be randomly allocated for normothermia therapy. Treatment will be initiated within 6 hours of the event, the child will be dressed with a cooling suit and their temperature will be monitored. Cooling will be to 36-37 °C . Treatment period will be 72 hrs.
  Interventions: Device: Whole body hypothermia
- Control (No Intervention): A group of children that underwent a cardiac surgery and was not suspected to have an hypoxic ischemic brain injury. This group will be undergo the similar biomarkers collection as arm 1 and 2. The information will be used to measure the change in biomarkers between surgeries with no HII to those in arm 1+2.

INTERVENTIONS:
Device: Whole body hypothermia — Treatment will be initiated within 6 hours of the event, the child will be dressed with a cooling suit and their temperature will be monitored. Cooling will be to 33 +/- 1 °C . Treatment period will be 48 hours with 24 hours warming up period.
  Other Names: ThermoWrap® cover and Alon® Control Unit
  Arms: Whole body hypothermia; Whole body normothermia

SUMMARY:
Cardiac pathology is a major risk for brain injury and neurodevelopmental deficit. The most common cause of cardiac pathology is congenital heart defects (CHD) about 4-8/1000 live births a year. The most common etiology of the brain insult is hypoxic ischemic injury (HII) as result of hemodynamic instability in the perioperative period. Similar insults in adults with cardiac arrest or infants with neonatal asphyxia, was successfully treated with hypothermia, initiated within 6 hours after the event. Although, hypothermia is most likely an effective treatment for HII in children with cardiac anomaly, it also carries a risk for bleeding or infection of the surgical wound. In this randomized control trial, hypothermia treatment will be compared to normothermia treatment of patients in the pediatric cardiac intensive care unit (PCICU) following severe HII in the PCICU or operating room. The effect will be quantified by MRI, serum biomarkers of brain injury, amplitude integrated EEG, neurological evaluation coagulation and infection evaluation in the acute phase and by developmental assessment at 1, 6 months and 2, 5 years. Favorable effect of hypothermia with minimal risks may open the door for the implementation of hypothermia as a standard care in PCICUs.

ELIGIBILITY:
Inclusion Criteria:

1. Every child entering the PCICU, age < 7 years
2. The child will enter arm 1 or 2 if he underwent the event described in section 3.
3. Hypoxic ischemic event that would render hypothermia treatment is defined as

   * During the hospitalization in the PCICU before or after the surgery:

   Resuscitation comprised of chest compressions for more than 2 minutes, and the first blood tests immediately after the resuscitation show a serum lactate level of more than 90 mg/dl OR Resuscitation comprised of chest compressions for more than 2 minutes, and the first blood tests immediately after the resuscitation shows a serum lactate level of more than 40 mg/dl and a blood pH level of less than 7.1
   * During the surgery Near infra red spectroscopy lower than 40 for more than 5 minutes AND Serum lactate levels of more than 90 mg/dl during the event OR The patient is re-connected to cardio-pulmonary bypass machine as a result of the event
4. Initiation of hypothermia treatment within 6 hours following the hypoxic ischemic event defined in section 3.

Exclusion criteria

* Suspected hypoxic ischemic event as described in the Inclusion Criteria in the 2 weeks prior to the PCICU admission
* Prolonged low cerebral perfusion before the PCICU admission, with 3 repeated tests in 1 hour of lactate level higher than 40 mg/dl and pH lower than 7.1
* Rejection criteria
* A second resuscitation after the hypoxic ischemic event and before a brain MRI is done

Ages: 1 Day to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Biomarkers | 48 hours after the surgery
  Each child will have 4 blood samples for biomarkers including S100B, Glial Fibrillary Acidic Protein and Specific Neuronal Enolase at the following schedule: before the cardiac surgery, within 6 hr after the surgery, 24 and 48 hrs after the surgery
Magnetic Resonance Imaging | 10 days after
  In arms 1 and 2 an MRI with the sequences of T1, T2, Diffusion Weighted Imaging, Diffuse Tensor Imaging and Magnetic Resonance Spectroscopy
Neurological Evaluation | 1 week
  Neurological assessment will be done prior to the cardiac surgery and and one week (or earlier if the child will be fully recovered and discharged before) using standard neurological evaluation, pediatric stroke outcome measure

SECONDARY OUTCOMES:
Short term neuro-developmental outcome | 2 months
  Neurological assessment using standard neurological evaluation, pediatric stroke outcome measure and pediatric cerebral performance category
Short term neuro-developmental outcome | 5 yrs
  At 2 and 5 yrs after the hypothermia treatment a c. Vineland adaptive behavior scale (Vineland™-II) will be done

CONTACTS AND LOCATIONS:
Overall Officials: Omer B Bar Yosef, MD-PhD, Principal Investigator — Chain Sheba Medical Ceneter